CLINICAL TRIAL: NCT00700505
Title: A Study to Determine the Safety and Efficacy of a New Non-invasive Heating Garment to Reduce Urinary Hesitancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ThermaRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR-DM-001
Record Dates: First submitted 2008-06-11; First posted 2008-06-18 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Urinary Retention; Urinary Hesitancy Intermittent
Keywords: Benign Prostatic Hyperplasia; BPH; Benign Prostatic Hypertrophy; Urinary Retention; Shy Bladder; Urinary Hesitancy; Bashful Bladder; Paruresis
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Heating Garment (Experimental): FlowPants(R) Garment with Heating
  Interventions: Device: FlowPants(R) Garment

INTERVENTIONS:
Device: FlowPants(R) Garment — The garment is shaped like a pair of boxer briefs. Garment heating is battery-powered.
  The garment is activated and begins to heat up 5-15 minutes prior to voiding.

SUMMARY:
To determine the safety and efficacy of the ThermaRx heating device for the application of controlled low level heat to improve symptoms of LUT dysfunction (hesitancy, urgency).

DETAILED DESCRIPTION:
This study will assess the safety and efficacy of ThermaRx heat treatment in subjects who have urinary hesitancy.

The rationale for this approach is based on anecdotal evidence and case reports suggesting that urinary hesitancy can be effectively reduced by external skin heating (hot tub "Jacuzzi" effect, perineal hot water spray). However, to date, there have been no formal studies of this non-invasive form of treatment, and the mechanism of action is still unclear.

This is a two-day study in which each subject will receive an oral fluid load and then one (1) heating treatment with the device. Ultrasound-based measurements of bladder volume will be performed both before and after voiding. On Day 1, voiding will be performed in a standing position; on Day 2, voiding will be done in a sitting position.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects 25-80 years of age at the screening visit.
* Subject must have mild-to-moderate urinary hesitancy symptoms (shown as an American Urological Association Symptom Index (AUA-SI) score of 7-19).
* Symptoms include (not limited to):
* Leaking or dribbling of urine
* More frequent urination, especially at night
* Urgency to urinate
* Urine retention (inability to urinate)
* Hesitant, interrupter or weak stream of urine
* Inability or difficulty to urinate in public

Exclusion Criteria:

* History of prostate cancer or prostate surgery
* Currently (or within the past 30 days) on active treatment for prostate problems

Ages: 25 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Post-void residual urinary volume (PVR) | Both Study Day 1 & 2 before/after oral fluid load

SECONDARY OUTCOMES:
Voided volume percentage (%) based on pre-void and post-void ultrasound volumes | Both Study Day 1 & 2 before/after oral fluid load

CONTACTS AND LOCATIONS:
Overall Officials: David Mobley, M.D., Principal Investigator — Mobley Clinical Research Center; John T La, Study Director — Mobley Clinical Research Center
Locations (1):
- Mobley Clinical Research Center, Houston, Texas, United States

REFERENCES:
- See also: Heat Therapy — http://www.thermarx.com